CLINICAL TRIAL: NCT04608123
Title: Effect of Bilateral Subthalamic Nucleus Deep Brain Stimulation on Neuropsychiatric Fluctuations in Patients With Parkinson's Disease, Evaluated With a New, Dedicated Scale
Brief Title: Effect of Deep Brain Stimulation on Neuropsychiatric Fluctuations in Patients With Parkinson's Disease
Acronym: PSYCHOSTIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 0
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease (Disorder)
Keywords: DBS; Deep Brain Stimulation; Neuropsychiatric Fluctuations; Nonmotor Fluctuations; Scale
MeSH Terms: conditions — Parkinson Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DBS Patients with NFS: Patients with PD treated with STN DBS between 2016 and 2019 who underwent NFS testing in pre and post-op conditions
  Interventions: Other: none (observational study)

INTERVENTIONS:
Other: none (observational study) — DBS

SUMMARY:
Retrospective, monocentric, observational study designed to evaluate the effects of Bilateral Subthalamic Nucleus Deep Brain Stimulation (DBS STN) on Neuropsychiatric fluctuations in Patients with Parkinson's Disease (PD)

DETAILED DESCRIPTION:
Pre-operative versus 12-Month Follow-Up analysis of changing in Neuropsychiatric Fluctuations Scale (NFS) score in preoperative versus postoperative MED OFF (during acute withdrawal of dopaminergic therapy) and MED ON (during super-liminal Levodopa dose) conditions. Postoperative evaluations are always performed with DBS turned on and stimulating (STIM ON)

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Treatment with Bilateral STN DBS
* Evaluation with NFS in both preoperative and 12 months post-surgery follow-up context

Exclusion Criteria:

* DBS for non PD patients
* Unilateral DBS or other DBS targets
* Patients not evaluated with NFS
* Patients with incomplete preoperative evaluation
* Patients who refused the use of their data

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: PD patients treated with DBS STN at Grenoble Hospital within September 2016 and June 2019
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness of DBS for Neuropsychiatric Fluctuations | 12 months after surgery
  Improvement of Neuropsychiatric Fluctuation Scale (NFS) Score between preoperative MED ON and MED OFF conditions versus postoperative MED ON-STIM ON and MED OFF-STIM ON conditions. NFS ON and OFF med scores are independent and they ranges from -30 to +30. Positive scores represent good outcomes (good feelings, non OFF neuropsychiatric symptoms), whereas negative scores denote the presence of negative feelings in a quantity exceeding the positive ones

SECONDARY OUTCOMES:
Preoperative and Postoperative demographical and clinical factors linked to a post-surgical change in Neuropsychiatric Fluctuations | 12 months
  Changing in pre-post op NFS scores correlated with:
  * Demographic and Clinical data: age, sex, disease duration, side onset, clinical phenotype, years passed with fluctuations, comorbidities, psychiatric history not linked to the disease or its treatment, psychiatric complications of dopaminergic therapy
  * Dopaminergic treatment data: years of therapy with Levodopa, percentage of motor improvement with Levodopa-test, pre and postoperative LEDD, changing in psychiatric treatment (doses and number of medications)
  * Perioperative variables: type of anaesthesia, perioperative complications
  * DBS parameters: stimulation type, plots selected, amplitude, rate, duration of impulse, stereo tactical coordinates of electrodes, stimulator type (rechargeable, not rechargeable)
Neuropsychiatric Fluctuations, Cognitive and Psychiatric state | 12 months
  Changing in pre-postop NFS scores correlated with:
  * Cognitive evaluation scales (Mattis Scale, Score Frontal, Wisconsin Card Sorting Test - WCST, Luria manual sequencing task)
  * Psychiatric evaluation scales (Beck Depression Scale - BDI-II, Evaluation Comportamentale dans la Maladie de Parkinson - ECMP, Starkstein Apathy Scale)
Neuropsychiatric Fluctuations, preoperative and postoperative motor status | 12 months
  Changing in pre-postop NFS scores correlated with:
  * Preoperative UPDRS III Score (total score, sub scores of tremor, rigidity, akinesia, parole, posture-gait-instability) in MED ON and MED OFF conditions
  * Changing in UPDRS III Scores (total and sub scores) in preoperative MED ON and MED OFF conditions versus postoperative MED ON STIM ON and MED OFF STIM ON conditions
Neuropsychiatric Fluctuations and other Nonmotor Symptoms | 12 months
  Changing in pre-postop NFS scores correlated with:
  - Changing in MDS-UPDRS scores and sub scores (total, section I, section II, section IV)
Neuropsychiatric Fluctuations and Dopaminergic Therapy | 12 Months
  Changing in pre-postop NFS scores correlated with:
  - Preoperative versus postoperative Levodopa equivalent dose (LEDD)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Moro, Study Director — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmitt E, Krack P, Castrioto A, Klinger H, Bichon A, Lhommee E, Pelissier P, Fraix V, Thobois S, Moro E, Martinez-Martin P. The Neuropsychiatric Fluctuations Scale for Parkinson's Disease: A Pilot Study. Mov Disord Clin Pract. 2018 Mar 23;5(3):265-272. doi: 10.1002/mdc3.12607. eCollection 2018 May-Jun. PMID 30363450
- [Result] Abbes M, Lhommee E, Thobois S, Klinger H, Schmitt E, Bichon A, Castrioto A, Xie J, Fraix V, Kistner A, Pelissier P, Seigneuret E, Chabardes S, Mertens P, Broussolle E, Moro E, Krack P. Subthalamic stimulation and neuropsychiatric symptoms in Parkinson's disease: results from a long-term follow-up cohort study. J Neurol Neurosurg Psychiatry. 2018 Aug;89(8):836-843. doi: 10.1136/jnnp-2017-316373. Epub 2018 Feb 7. PMID 29436490
- [Result] Hogg E, Wertheimer J, Graner S, Tagliati M. Deep Brain Stimulation and Nonmotor Symptoms. Int Rev Neurobiol. 2017;134:1045-1089. doi: 10.1016/bs.irn.2017.05.022. Epub 2017 Jul 3. PMID 28805564
- [Result] Kurtis MM, Rajah T, Delgado LF, Dafsari HS. The effect of deep brain stimulation on the non-motor symptoms of Parkinson's disease: a critical review of the current evidence. NPJ Parkinsons Dis. 2017 Jan 12;3:16024. doi: 10.1038/npjparkd.2016.24. eCollection 2017. PMID 28725706
- [Result] Azulay JP, Witjas T, Eusebio A. Effect of subthalamic deep brain stimulation on non-motor fluctuations in Parkinson's disease. J Neural Transm (Vienna). 2013 Apr;120(4):655-7. doi: 10.1007/s00702-012-0958-9. Epub 2012 Dec 23. PMID 23263599